CLINICAL TRIAL: NCT04285359
Title: Impact of Severe Intraoperative Hyperglycemia on Infection Rate After Elective Intracranial Interventions
Status: Completed | Type: Observational
Sponsor: Burdenko Neurosurgery Institute (Other)
Responsible Party: Sponsor
Other Study IDs: PPN-2020-02-06
Record Dates: First submitted 2020-02-22; First posted 2020-02-26 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2020-10

CONDITIONS: Hyperglycemia; Craniotomy; Infection Post Op
MeSH Terms: conditions — Hyperglycemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Intracranial Interventions — Neurosurgical elective intracranial interventions: supra- and infratentorial craniotomies, transnasal endoscopic interventions.

SUMMARY:
Severe intraoperative hyperglycemia (SIH) is recognized as one of the important risk factors for the increasing of the postoperative infections rate, which can negatively affect the final outcome of surgical treatment. Studies in recent years have shown a much higher incidence of wound infections, respiratory and urinary tract infections in patients who intraoperatively had an increase in blood glucose level (BGL) above 180 mg/dl (10 mmol/l). This problem in neurosurgery is especially important due to the high proportion of patients with acute injuries and potentially long-term need for postoperative intensive care, as well as the frequent use of drugs that increase blood glucose level (steroids) in neurooncology. Most published studies include patients from both of these groups. This study is aimed to assess the impact of severe intraoperative hyperglycemia on the incidence of infectious complications only in patients scheduled for elective intracranial interventions.

ELIGIBILITY:
Inclusion Criteria:

Adult patients (>18 years) scheduled for elective intracranial (open or endoscopic) intervention.

Exclusion Criteria:

Diagnosis of infection (local or systemic) in preoperative period; urgent intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 years) scheduled for elective intracranial intervention.
Sampling Method: Probability Sample
Enrollment: 514 (Actual)
Dates: Start 2020-10-28 (Actual); Primary Completion 2021-03-15 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Infection rate | 7 days after surgery
  Proportion of patients diagnosed with infection (wound, pulmonary, urological, blood etc.) in the postoperative period according to CDC.

SECONDARY OUTCOMES:
Antibiotic prophylaxis | Preoperatively
  Antibiotic usage for prevention of postop infection: type and dosage
Glucose level | Twice intraoperatively: before incision and at the end of surgery
  Intraoperative glucose level in whole blood
History of steroids usage | Preoperatively
  Dosages and regimen of dexamethasone in the perioperative period
Insulin dosage | Intraoperatively
  Intraoperative dose of insulin
Complications | Intraoperatively
  Perioperative complications (episodes of hemodynamic instability, blood loss, etc.)
Duration of stay in ICU and hospital | 30 days
  Length of stay in ICU (in hours) and in hospital (in days) after surgical intervention
Treatment outcome | 30 days
  Outcome at the moment of discharge (improved,unchanged, worsened, death)

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Kulikov, Principal Investigator — Burdenko National Medical Research Center of Neurosurgery
Locations (2):
- Sapienza University of Rome, Roma, Italy
- Federal State Autonomous Institution "N .N. Burdenko National Medical Research Center of Neurosurgery" of the Ministry of Healthcare of the Russian Federation, Moscow, Russia

REFERENCES:
- [Derived] Kulikov A, Krovko Y, Nikitin A, Shmigelsky A, Zagidullin T, Ershova O, Gadzhieva O, Bilotta F. Severe Intraoperative Hyperglycemia and Infectious Complications After Elective Brain Neurosurgical Procedures: Prospective Observational Study. Anesth Analg. 2022 Nov 1;135(5):1082-1088. doi: 10.1213/ANE.0000000000005912. Epub 2022 Jan 20. PMID 35051950